CLINICAL TRIAL: NCT01500850
Title: Establishing Cardiovascular Biomarkers to Define Preferred Lantus® Use.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ikfe-CRO GmbH (Industry)
Collaborators: IKFE Institute for Clinical Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lantu_L_05720
Record Dates: First submitted 2011-12-05; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Insulin-requiring Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes mellitus; NPH insulin; Insulin Glargine; cardiovascular biomarkers; hsCRP, adiponectin; intact proinsulin; cardiovascular risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin, Isophane; Insulin; Insulin Glargine; insulin glulisine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- NPH insulin + insulin glulisine (Active Comparator): Patients will be randomized to be treated with NPH insulin + Insulin Glulisine for 24 weeks.
  Interventions: Drug: nph insulin; Drug: Insulin glulisine
- NPH insulin + human insulin (Active Comparator): Patients will be randomized to be treated with NPH insulin + human insulin for 24 weeks.
  Interventions: Drug: human insulin
- Insulin glargine + insulin glulisine (Experimental): Patients will be randomized to be treated with insulin glargine + insulin glulisine for 24 weeks.
  Interventions: Drug: Insulin Glargine; Drug: Insulin glulisine
- Insulin Glargine + Human insulin (Experimental): Patients will be randomized to be treated with insulin glargine + human insulin for 24 weeks.
  Interventions: Drug: human insulin; Drug: Insulin Glargine

INTERVENTIONS:
Drug: nph insulin — Dosage will be pro re nata. Patients should aim an blood glucose level of ≤ 100 mg/dL.
  Other Names: Insuman Basal
  Arms: NPH insulin + insulin glulisine
Drug: human insulin — Dosage will be pro re nata. Patients should aim an blood glucose level of ≤ 100 mg/dL.
  human insulin: bolus injections before each main meal
  Other Names: Insuman Rapid
  Arms: Insulin Glargine + Human insulin; NPH insulin + human insulin
Drug: Insulin Glargine — Dosage will be pro re nata. Patients should aim an blood glucose level of ≤ 100 mg/dL.
  Other Names: Lantus
  Arms: Insulin Glargine + Human insulin; Insulin glargine + insulin glulisine
Drug: Insulin glulisine — Dosage will be pro re nata. Patients should aim an blood glucose level of ≤ 100 mg/dL.
  Insulin glulisine: bolus injections before each main meal
  Other Names: Apidra
  Arms: Insulin glargine + insulin glulisine; NPH insulin + insulin glulisine

SUMMARY:
The aim of this study is to observe changes in cardiovascular biomarkers during treatment with Lantus in patients with Type 2 Diabetes mellitus.

DETAILED DESCRIPTION:
* Phase IV
* Indication: Diabetes mellitus Type 2
* Primary objective:

To compare fasting intact proinsulin secretion at the beginning and after a 24 week treatment period.

- Secondary objectives: To evaluate changes in the parameters

* insulin,
* glucose,
* intact proinsulin (after a glucose challenge),
* hsCRP,
* adiponectin,
* MMP-9,
* HbA1c,
* weight

after 24 weeks of treatment.

To investigate the changes of

* glucose,
* intact proinsulin,
* hsCRP,
* adiponectin,
* HbA1c
* weight

between visit 2 (baseline), visit 6 (12 weeks) and visit 8 (final visit after 24 weeks).

To investigate the number of patients with normal values for parameters hsCRP, adiponectin, and intact proinsulin after 24 weeks of treatment (responder rates).

-Primary efficacy variable: Fasting intact proinsulin concentration at timepoint Visit 2 (Baseline) and Visit 8 (after 24 week treatment)

-Secondary efficacy variables: All secondary parameters will be assessed after 24 weeks of treatment and compared versus baseline assessment.

* Weight
* hsCRP
* Adiponectin
* MMP-9
* OGTT parameters (insulin, intact proinsulin, glucose at time point 0, 60 and 120 minutes after 24 weeks
* HOMA-IR score
* HbA1c

Additionally the following parameters will be assessed at visit 6 and will be compared with visit 2 and visit 8:

* Weight
* hsCRP
* Adiponectin
* Fasting intact Proinsulin
* Glucose
* HbA1c
* Safety Variables:
* Adverse Events
* Hypoglycaemic events

Medication/Dosage:

Insulin glargine, dose individually adapted to reach treatment goal (FBG ≤ 100 mg/dL)NPH Insulin, dose individually adapted to reach treatment goal (FBG ≤ 100 mg/dL)Insulin glulisine, dose individually adapted to reach treatment goal (FBG ≤ 100 mg/dL)Human Insulin, dose individually adapted to reach treatment goal (FBG ≤ 100 mg/dL)

-Study Duration: Duration of study participation for one patient is approximately 26 weeks. Overall total duration of the study is approximately 10 months.

Design:

This is a randomized in four arms, open-label, multi-center study. Population Patients with Type 2 Diabetes mellitus, Sample Size n = 60 (15 per arm)

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent.
* Patient consents that his/her family physician/diabetologist will be informed of trial participation
* Type-2 diabetes mellitus ≥ 1 year of diagnosis (male and female)
* Experienced in self blood glucose measurement for ≥ 3 months.
* HbA1c ≤ 9% and >6,5%
* BMI > 30 kg/m²
* Age ≥ 18 years
* Waist circumference > 88 cm (female) and > 102 cm (male)
* NPH insulin treatment plus 1 or 2 OAD (except TZD)

Exclusion Criteria:

* History of drug or alcohol abuse within the last five years prior to screening
* Anamnestic history of hypersensitivity to the study drugs (or any component of the study drug) or to drugs with similar chemical structures
* History of severe or multiple allergies
* Treatment with any other investigational drug within 3 months prior to screening
* Progressive fatal disease
* History of significant cardiovascular, respiratory, gastrointestinal, hepatic (ALAT and/or ASAT > 3 times the normal reference range), renal (creatinine > 1.3 mg/dl in women and >1.6 mg/dl in men), neurological, psychiatric and/or hematological disease as judged by the investigator
* Pregnant or lactating women
* Sexually active women of childbearing potential not consistently and correctly practicing birth control by implants, injectables, combined oral contraceptives, hormonal intrauterine devices (IUDs), sexual abstinence or vasectomized partner
* Treatment with GLP1-analog or Thiazolidinediones (TZD)
* hsCRP > 10 mg/l (by rapid test at screening visit).
* Lack of compliance or other similar reason that, according to investigator, precludes satisfactory participation in the study
* Type 1 Diabetes mellitus
* Patients already treated with intensified conventional insulin therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Fasting Intact Proinsulin | Change from baseline at 24 weeks
  The difference of fasting intact proinsulin after 24 weeks of treatment compared to baseline.

SECONDARY OUTCOMES:
Weight | Baseline and after 24 weeks of treatment.
  To evaluate the changes of weight after 24 weeks of treatment compared to baseline.
hsCRP | Baseline and after 24 weeks of treatment.
  To evaluate changes of hsCRP after 24 weeks of treatment compared to baseline.
Adiponectin | Baseline and after 24 weeks of treatment.
  To evaluate changes of adiponectin after 24 weeks of treatment compared to baseline.
MMP-9 | Baseline and after 24 weeks of treatment.
  To evaluate changes of MMP-9 after 24 weeks of treatment compared to baseline.
OGTT parameters (insulin, intact proinsulin, glucose at time point 0, 60 and 120 minutes after 24 weeks | Baseline and after 24 weeks of treatment.
  To evaluate changes of OGTT parameters (insulin, intact proinsulin, glucose at time point 0, 60 and 120 minutes) after 24 weeks of treatment compared to baseline.
HOMA-IR score | Baseline and after 24 weeks of treatment.
  To evaluate changes of HOMA-IR score after 24 weeks of treatment compared to baseline.
HbA1c | Baseline and after 24 weeks of treatment.
  To evaluate changes of HbA1C after 24 weeks of treatment compared to baseline.
Weight | After 12 weeks of treatment compared to baseline and to 24 weeks of treatment.
  To evaluate changes of weight after 12 weeks of treatment compared to baseline and compared to 24 weeks.
hsCRP | After 12 weeks of treatment compared to baseline and to 24 weeks of treatment.
  To evaluate changes of hsCRP after 12 weeks of treatment compared to baseline and compared to 24 weeks.
Adiponectin | After 12 weeks of treatment compared to baseline and to 24 weeks of treatment.
  To evaluate changes of adiponectin after 12 weeks of treatment compared to baseline and compared to 24 weeks.
Fasting intact Proinsulin | After 12 weeks of treatment compared to baseline and to 24 weeks of treatment.
  To evaluate changes of fasting intact proinsulin after 12 weeks of treatment compared to baseline and compared to 24 weeks.
Glucose | After 12 weeks of treatment compared to baseline and to 24 weeks of treatment.
  To evaluate changes of Glucose after 12 weeks of treatment compared to baseline and compared to 24 weeks.
HbA1c | After 12 weeks of treatment compared to baseline and to 24 weeks of treatment.
  To evaluate changes of HbA1c after 12 weeks of treatment compared to baseline and compared to 24 weeks.
Responder rate | After 24 weeks of treatment compared to baseline.
  To investigate the number of patients with normal values for parameters hsCRP, adiponectin, and intact proinsulin after 24 weeks of treatment (responder rates).
Hypoglycemic events. | Baseline up to 24 weeks.
  Hypoglycemic events defined as blood glucose below 63 mg/dl.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Pfützner, Professor, Principal Investigator — Ikfe GmbH
Locations (1):
- ikfe GmbH, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419